CLINICAL TRIAL: NCT02873637
Title: Adductor Under Sartorial Canal Catheter (KTT) Versus Femoral Catheter (KTF) in a Quick Rehabilitation Process After Total Knee Replacement: A Controlled, Randomized Study (KTSS)
Brief Title: Adductor Under Sartorial Canal Catheter (KTT) Versus Femoral Catheter (KTF) in a Quick Rehabilitation Process After Total Knee Replacement
Acronym: KTSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHD050-16
Record Dates: First submitted 2016-08-12; First posted 2016-08-19 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Total Knee Replacement
Keywords: total knee replacement; anesthesia; catheter

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- under sartorial catheter (Experimental): catheter under sartorial
  Interventions: Device: under sartorial catheter
- femoral catheter (Other): femoral catheter
  Interventions: Device: femoral catheter

INTERVENTIONS:
Device: under sartorial catheter
  Arms: under sartorial catheter
Device: femoral catheter
  Arms: femoral catheter

SUMMARY:
The main objective of this study is to show that postoperative Total Knee Replacement (TKR), an analgesic perineural catheter in position under sartorial (KTSS) best preserves motor quadriceps femoral perineural catheter that (KTF) infused with even low doses of local anesthetics, this motor being evaluated by a semi quantitative simple clinical test locking of the knee feasible at the bedside.

Patients will be randomized in two arms:

* catheter in position under sartorial (experimental group)
* femoral catheter (control group)

ELIGIBILITY:
Inclusion Criteria:

* Major Patient (≥ 18 years)
* Before tricompartmental benefit from knee replacement (TKR) unilateral,
* TKR programmed on one of the first three days of the week (Monday to Wednesday)
* Physical status score I-III,
* Non septic programmed surgery under general anesthesia
* Able to understand the protocol
* Written informed consent
* Social Insured
* Opportunity to be followed under the Protocol

Exclusion Criteria:

* Age ≥ 85 years
* Obesity (BMI ≥ 35)
* Revision TKR,
* Patients not cooperating or not including the French,
* Difficulties in understanding and evaluating the score pain (VAS),
* Preoperative cognitive dysfunction making unreliable interrogation
* Patient unable to read and / or write (literacy, ...)
* Known bleeding disorders,
* Vascular surgery for femoral vessels on the operated side,
* Neuropathy of the lower limb,
* Localized infection at the puncture catheters,
* Known allergy to ropivacaine,
* Renal and / or severe hepatic impairment,
* Taking opioids for more than a month before surgery,
* Intolerance to morphine,
* Rheumatic inflammatory disease,
* Patients receiving immunosuppressive therapy or long-term corticosteroid
* Allergy or against-indications to standard treatments administered intraoperative and postoperative
* Flexion deformity> 10 ° or valgus deformity with significant
* Refused to participate
* Patient trusteeship, guardianship, deprived of liberty
* Women premenopausal who become pregnant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-11-11 (Actual)

PRIMARY OUTCOMES:
International clinical score Daniels and Worthingham | 2 day after surgery (total knee replacement)
  This score measures the driving force of the quadriceps (scale M0: no contraction in M5: normal force)

CONTACTS AND LOCATIONS:
Locations (1):
- CHD Vendée de la Roche sur Yon, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guilley J, Besancon I, Hivert A, Plouhinec AM, Oudot M, Venet G, Fraquet N, Cousin J, Planche L, Ganiere C, Duchalais A. Femoral nerve inguinal approach versus proximal femoral triangle ap proach for continuous regional analgesia in active rehabilitation after total knee arthroplasty: A prospective, randomised study. Anaesth Crit Care Pain Med. 2022 Apr;41(2):101043. doi: 10.1016/j.accpm.2022.101043. Epub 2022 Feb 19. PMID 35189397